CLINICAL TRIAL: NCT06246331
Title: An Observational Study on the Clinical Efficacy and Safety of BriTurn Injection or BrisTurn Prefilled Injection Administered for Reversal of Neuromuscular Blockade in Patients Receiving General Anesthesia
Brief Title: Evaluation of the Clinical Efficacy and Safety of BriTurn Injection or BrisTurn Prefilled Injection
Status: Recruiting | Type: Observational
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-BRT-401
Record Dates: First submitted 2023-12-20; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Reversal of Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluate clinical efficacy and safety in adult patients administered BriTurn injection or BrisTurn Prefilled injection for reversal of neuromuscular blockade induced by Rocuronium or Vecuronium.

DETAILED DESCRIPTION:
This study evaluate clinical efficacy and safety in adult patients administered BriTurn injection or BrisTurn Prefilled injection for reversal of neuromuscular blockade induced by Rocuronium or Vecuronium.

* Efficacy: Time (minutes) for Train-Of-Four (TOF) ratio to reach 0.9 (90%)
* Safety: whether bradycardia and resulting cardiac arrest occur or whether bronchospasm occurs

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years of age
* Subject administered BriTurn Injection or BrisTurn Prefilled Injection for reversal of neuromuscular blockade induced by Rocuronium or Vecuronium

Exclusion Criteria:

* Pregnant women or nursing women
* Subject to prohibition according to the permission of BriTurn Injection or BrisTurn Prefilled Injection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 19 years or older
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time (minutes) for Train-Of-Four (TOF) ratio to reach 0.9 (90%) | after administration of BriTurn Injection or BrisTurn Prefilled Injection up to 3 minutes
  Time (minutes) for Train-Of-Four (TOF) ratio to reach 0.9 (90%) after administration of BriTurn Injection or BrisTurn Prefilled Injection up to 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sangseok Lee, Principal Investigator — Inje University
Locations (1):
- Inje University Sanggye Paik Hospital, Seoul, South Korea